CLINICAL TRIAL: NCT01325246
Title: Correlation Between Reoperation and Clinical Palpable Recurrence 3 Years After Ventral Hernia Repair
Brief Title: Reoperation Rate Versus Clinical Recurrence After Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: FH-1
Record Dates: First submitted 2010-09-14; First posted 2011-03-29 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Ventral Hernia
Keywords: ventral hernia; repair; clinical; reoperation
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The risk for recurrence after ventral hernia repair is often based on reoperation rates with short follow-up rather than recurrences identified by clinical examinations.

The purpose of current study is find the real incidence of recurrences 3 years after ventral hernia repair and to compare with the reoperation rate.

DETAILED DESCRIPTION:
all patients in a restricted area (all patients in the part of Denmark called Zealand) who had a ventral hernia repair in 2007 (appr. 1200 patients). The patients will be sorted by a questionnaire and if the patients are suspicious for recurrence they will be offered a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Primary ventral hernia repair performed in the region of Zealand in Denmark

Exclusion Criteria:

* Patients who died and patients not resident in region Zealand

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1200 patients who had a ventral hernia repair in 2007
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Clinical recurrence after ventral hernia repair | up to 4 years

SECONDARY OUTCOMES:
explanations for not having a recurrence repair | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — dept. of surgery, Køge Hospital
Locations (1):
- Dept. of surgery, Køge Hospital, Køge, Denmark

REFERENCES:
- [Derived] Helgstrand F, Rosenberg J, Kehlet H, Strandfelt P, Bisgaard T. Reoperation versus clinical recurrence rate after ventral hernia repair. Ann Surg. 2012 Dec;256(6):955-8. doi: 10.1097/SLA.0b013e318254f5b9. PMID 22580941